CLINICAL TRIAL: NCT04999631
Title: Neoadjuvant Squaric Acid Dibutylester Treatment of Melanocytes in Congenital Melanocytic Nevi
Brief Title: SADBE for Congenital Melanocytic Nevi
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elena Hawryluk, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMN001
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Congenital Melanocytic Nevus
MeSH Terms: interventions — squaric acid dibutyl ester

STUDY DESIGN:
Intervention Model Description: Two areas of the subject's nevus will be marked. Study medication will be applied to one area. Placebo ethanol solution will be applied to the other area. Area to be treated will be randomized among subjects. Both areas will be monitored and following surgery, samples will be obtained. Area to be treated vs area that will serve as control will be randomized.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded on what area received the study cream and what area received the placebo ethanol solution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Squaric Acid Dibutyl Ester (SADBE) (Experimental): Following sensitization, subjects will apply 0.2% SADBE in ethanol to a predetermined area of their nevus 3 times per week for 12 weeks, with adjustment of frequency depending on response.
  Interventions: Drug: Squaric Acid Dibutyl Ester
- Control (Placebo Comparator): Subject will apply an ethanol solution to a specified area of the nevus.
  Interventions: Drug: Ethanol Solution

INTERVENTIONS:
Drug: Squaric Acid Dibutyl Ester — Topical squaric acid dibutyl ester (SADBE) dissolved in ethanol at 0.2% concentration.
  Arms: Squaric Acid Dibutyl Ester (SADBE)
Drug: Ethanol Solution — Control
  Arms: Control

SUMMARY:
A study to evaluate the safety and efficacy topical squaric acid dibutylester (SADBE) for the neoadjuvant treatment of congenital melanocytic nevi (CMN).

DETAILED DESCRIPTION:
Patients with CMN and plans for elective surgical resection of their nevi will be enrolled in the study. Two clinically similar areas within the planned excision site will be identified, marked and treated with SADBE or the placebo solution. Following surgical resection, samples from the excised nevi will be taken and assessed for number of melanocytes. Incidence of adverse events will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Subject or parents willing and able to give informed consent, and assent as appropriate.
* Patients who have a clinical diagnosis of CMN with plans for elective non-urgent excision of part or all of their nevus, with nevus surface area of > 6 cm2.

Exclusion Criteria:

* Immunosuppressive therapy with glucocorticoid or other systemic immunosuppressant within 4 weeks of recruitment (except for inhaled corticosteroids for asthma).
* History of malignancy.
* History of organ transplantation.
* Known immunosuppressive disease, including infection with HIV.
* Severe medical comorbidities (diabetes mellitus requiring insulin, CHF of any severity, MI, CVA, or TIA within 3 months of screening visit, unstable angina pectoris, oxygen-dependent severe pulmonary disease)
* Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
* Subjects who have known hypersensitivity to SADBE or any of its components.
* Any condition judged by the investigator to cause this clinical trial to be detrimental to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of melanocytes per mm2 | 12 weeks
  The number of melanocytes present in the biopsy specimen will be measured. b. Assessment of pigment within stratum corneum, epidermis, and dermis

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 weeks
  The frequency of adverse events from each treatment arm will be compared.

OTHER OUTCOMES:
Clinical appearance of nevi | 12 weeks
  Treated areas will be compared for pigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Elena B. Hawryluk, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No